CLINICAL TRIAL: NCT05773378
Title: Do Intravaginal Devices Reduce or Eliminate Exercise Induced Urinary Incontinence in Female Runners?
Brief Title: Do Intravaginal Devices Reduce Urinary Incontinence in Female Runners?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Linda McLean, Professor in the School of Rehabilitation Sciences at University of Ottawa, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-06-22-8219
Record Dates: First submitted 2023-01-14; First posted 2023-03-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Urinary Incontinence
Keywords: exercise-induced urinary incontinence; running-induced urinary incontinence; intravaginal pessary; tampon; pelvic floor
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pessary Intervention (Experimental): Participants randomized to this group will receive an Uresta Incontinence Pessary to use each time they run over a 10-week period. They will be instructed to use the pessary only while running and remove it and wash it with soap and water when the training is over.
  Uresta is a reusable and removable device made of hypoallergenic medical-grade resin that is inserted into the vagina to provide mechanical support. It comes with a starter kit with 3 different sizes which work for over 80% of women. Participants will be instructed on how to test the 3 sizes to find out which one is right for them.
  Interventions: Device: Pessary Intervention
- Tampon Intervention (Experimental): Participants randomized to this group will receive 60 regular Tampax tampons and will be instructed to use them each time they run over a 10-week period. The tampon should be used only while running and removed and discarded when the training is over. Four weeks after the intervention (at the 16 weeks follow-up), they will receive a pessary with instruction how to use it if they desire so.
  Interventions: Device: Tampon Intervention
- Control Group (No Intervention): Participants randomized to this group won't receive any intervention and will be asked to continue their running training as usual for 10-weeks. They will also be instructed to not begin any treatment for urinary incontinence until their reassessment. Four weeks after the intervention (at the 16 weeks follow-up), they will receive a pessary with instruction how to use it if they desire so.

INTERVENTIONS:
Device: Pessary Intervention — Participants will receive a 3-size fitting kit and will fit the appropriate size based on manufacturer instruction. Once the size is verified, the participants will be asked to use the pessary while running over a 10-week period.
  Arms: Pessary Intervention
Device: Tampon Intervention — Participants will receive 60 regular Tampax tampons and will be instructed to use them each time they run over a 10-week period.
  Arms: Tampon Intervention

SUMMARY:
More than one in five females experience the embarrassment and shame of urine leakage while exercising and this urinary incontinence (UI) is a substantial barrier to exercise. As many as one in three females with UI report that they limit their physical activity due to incontinence: 11.6% by not exercising at all, 11.3% by exercising less and 12.4% by changing the type of exercise they perform. It is imperative to look for alternatives to manage this condition, as it is a key reason why females abandon the very physical exercise that is necessary to maintain or improve their physical and mental health and their quality of life.

While there is Grade A evidence for pelvic floor muscle training and some evidence for intravaginal pessaries to reduce symptoms of UI in general female populations, no study has evaluated the impact of conservative interventions specifically on UI experienced predominantly during running.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is a serious public health concern, imposing a significant financial burden. In Canada the direct and indirect health costs associated with UI total over 3.6 billion annually and no estimates of disease burden take into account deconditioning that results from withdrawal from physical activity nor effects on mental health or quality of life. Although the primary risk factor for UI is pregnancy and vaginal delivery, it was recently reported that between 20% and 40% of nulliparous females report urine leakage when they engage in physical activity.

Urinary continence is maintained as long as urethral closure pressure remains higher than bladder pressure. This is accomplished through a complex combination of mechanisms, including smooth and striated urethral sphincter muscle action, urethral venous engorgement and mucous secretions within the urethra, and the proper transfer of loads to the urethra, which depends on adequate bladder neck and urethral connective tissue support as well as pelvic floor muscle (PFM) action. The associations among physical activity, pelvic floor morphology and function, and UI are not clear. A recent systematic review retrieved 18 mainly small studies investigating the association between physical activity and pelvic floor dysfunction. Exercise at mild to moderate intensity appears to be protective, decreasing both the odds and the risk of experiencing urinary incontinence. However, females who engage in high-impact activities such as running are more likely to report UI during exercise than those who engage in mild or moderate intensity exercise, thus chronic and repetitive loading of the pelvic floor may have negative consequences.

While there is Grade A evidence for pelvic floor muscle training and some evidence for intravaginal pessaries to reduce symptoms of UI in general female populations, no study has investigated about interventions specific to running-induced UI.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years and over who run at least twice a week for a minimum of 10K/week (minimum speed of 6 km/h to ensure high impact), who have done so for at least 6 months (to ensure adequate duration of exposure), and who commit to continue the same amount during the study period
* Who regularly (≥ 1 per week) experience urine leakage while running.

Exclusion Criteria:

* Any risk factors related to exercise;
* Pain or musculoskeletal injury at the time of the screening;
* History of urogenital surgery;
* Symptoms of the female athlete triad;
* Have a known neurologic disorder (e.g. stroke, multiple sclerosis);
* Pregnancy or partum within the previous year;

For the in-lab assessment:

* Ability to run with a moderately full bladder for 38 minutes on a treadmill
* BMI ≥ 30
* Pelvic organ prolapse ≥ 2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Urinary leakage tracking: Proportion of training sessions during which urine leakage occurred | at baseline, and during intervention week 10-12
  At baseline, participants will be asked to complete a bladder diary, recording leakage experiences during each running session over a two-week period, while running without any intervention. This tracking will be repeated for another two-week period starting in the eighth week of running with the intervention (weeks 10-12 of the protocol). Participants will receive daily reminders to fill it out.
Patient's global impression of improvement | Post-intervention at 12 weeks, with follow-ups at 16, 24, and 36 weeks
  Participants will be asked to rate their overall impression of symptom improvement over the 10-week intervention on a 7 step scale (7= very much worse, to 1= very much better). Also, a follow-up will be conducted upon finishing the intervention, and, if they are still using the intervention, participants will be invited to rate their overall impression again at 16, 24 and 36 weeks.
Patient's global satisfaction with treatment | Post-intervention at 12 weeks, with follow-ups at 16, 24, and 36 weeks
  The participants will be asked how satisfied they were with their progress during the 10-weeks, on a scale from 0 to 100% (0 = not at all satisfied, 100 = completely satisfied). Also, a follow-up will be conducted upon finishing the intervention, and, if they are still using the intervention, participants will be invited to rate their satisfaction again at 16, 24 and 36 weeks.
International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms Modules (ICIQ-FLUTS) | Baseline, and post-intervention at 12 weeks, with follow-ups at 16, 24, and 36 weeks
  The ICIQ-FLUTS is a questionnaire for evaluating female lower urinary tract symptoms and impact on quality of life in research and clinical practice, with validity, reliability and responsiveness established with rigour in several data sets. It has a total of 12 questions; four questions on filling symptoms, three on voiding symptoms and five questions on urinary incontinence symptoms. The overall score ranges from 0-48, where all subscales scores are added. Higher scores indicate greater impact of individual symptoms for the patient.
  Participants will be asked to complete it at baseline and after 12-weeks. Also, a follow-up will be conducted upon finishing the intervention, and participants will be invited to complete the questionnaire again at 16, 24 and 36 weeks.
International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | Baseline, and post-intervention at 12 weeks, with follow-ups at 16, 24, and 36 weeks
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) is a questionnaire that includes three questions about urinary incontinence frequency, severity, and impact on daily life, resulting in a score of 0-21. The fourth question aims to classify the type of urinary incontinence, for this study 'leaks when you are physically active/exercising.' The questionnaire has a Level A validation grade according to ICI standards, as its validity, reliability, and responsiveness have been tested in several data sets. Participants will be asked to complete it at baseline and after 12-weeks. Also, a follow-up will be conducted upon finishing the intervention, and participants will be invited to complete the questionnaire again at 16, 24 and 36 weeks.

SECONDARY OUTCOMES:
Intervention questionnaire | Post-intervention at 12 weeks, with follow-ups at 16, 24, and 36 weeks
  A custom questionnaire with 20 questions was developed to collect information regarding participant's experience running with the intervention (tampon or pessary). The questions addresses the frequency of intervention use, ease of insertion and removal, comfort level while using the device, unintended effects (bleeding, vaginal discharge, pain), overall satisfaction, and the extent of urine leakage with the dispositive. Each question is rated on a scale form 0 to 100, with higher scores indicating a greater experience with the intervention. Participants randomized to the intervention groups will be asked to complete the questionnaire related to their assigned intervention after 12-weeks. Additionally, a follow-up will be conducted upon completing the intervention, and participants will be invited to complete the questionnaire again at 16, 24 and 36 weeks later.
Adherence to each intervention | Once a week during the 12 weeks of the study
  Adherence to the interventions will be logged through weekly e-mail and/or text contact, followed up with telephone contact if there is no response to the e-mail/text.
Unintended effects | Once a week during the 12 weeks of the study
  Adverse events (bleeding, vaginal discharge, pain, etc.) will be assessed through weekly e-mail/text contact, followed up with telephone contact if there is no response to the e-mail/text.
Brisk walking and Running lower Urinary Tract Symptoms Questionnaire (BRUTS) score | Baseline, and post-intervention at 12 weeks, with follow-ups at 16, 24, and 36 weeks
  The Brisk walking and Running Lower Urinary Tract Symptoms Questionnaire evaluates the symptoms and management strategies associated with urinary urgency and urinary incontinence that occurs during brisk walking, jogging, and running. Participants will be asked to complete it at baseline and post intervention (after 12-weeks). Also, a follow-up will be conducted upon finishing the intervention, and participants will be invited to complete the questionnaire again at 16, 24 and 36 weeks.
  The questionnaire has 4 domains: (1) about urgency symptoms, (2) about urgency urinary incontinence (UUI), (3) about stress urinary incontinence (SUI) and (4) about symptoms management. Scores are all 0-100 and higher scores mean a worse outcome with regards to the impact of lower urinary tract symptoms. The total score is still out of 100 (Urgency + UUI + SUI + Management / 4).
Changes in bladder neck height | Baseline and post intervention (at 12 weeks)
  A subgroup of participants will be invited for an in-lab assessment of pelvic floor morphology before and after running. Changes in bladder neck height will be assessed using ultrasound imaging at baseline and after 12 weeks. The images will be recorded before and after a 30-minute treadmill running protocol
Changes in levator hiatus area | Baseline and post intervention (at 12 weeks)
  A subgroup of participants will be invited for an in-lab assessment of pelvic floor morphology before and after running. Changes in levator hiatus area will be assessed by Ultrasound imaging at baseline and after 12-weeks. The images will be recorded before and after a 30-minute running protocol on a treadmill.
Changes in levator plate length | Baseline and post intervention ( at 12 weeks)
  A subgroup of participants will be invited for an in-lab assessment of pelvic floor morphology before and after running. Changes in levator plate lenght will be assessed by Ultrasound imaging at baseline and after 12-weeks. The images will be recorded before and after a 30-minute running protocol on a treadmill.
Changes in pelvic floor muscle strength | Baseline and post intervention ( at 12 weeks)
  A subgroup of participants will be invited for an in-lab assessment of pelvic floor morphology before and after running. Changes in pelvic floor muscle strength will be assessed at baseline and after 12-weeks using an intravaginal dynamometer. The measures will be recorded before and after a 30-minute running protocol on a treadmill.
Changes in pelvic floor muscle stiffness | Baseline and post intervention ( at 12 weeks)
  A subgroup of participants will be invited for an in-lab assessment of pelvic floor morphology before and after running. Changes in pelvic floor muscle stiffness will be assessed at baseline and after 12-weeks using an intravaginal dynamometer. The measures will be recorded before and after a 30-minute running protocol on a treadmill.
Pad weight gain | Baseline and post intervention ( at 12 weeks)
  A subgroup of participants will be invited for an in-lab assessment of pelvic floor morphology before and after running. These participants will be provided with a pre-weighed pad to attach to their underwear and wear it while running for 30 minutes on the treadmill. Once they finish running, the pad will be weighted again to record urine leakage. This will be done at the baseline and after 12-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Linda McLean, Principal Investigator — University of Ottawa
Locations (1):
- McLean Function Measurement Lab, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Spreadsheets will be provided by email upon request and based on the planned use of the data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 10 years after the publication of the study results.
Access Criteria: Planned use of data for systematic review or meta-analysis.

REFERENCES:
- [Background] Herschorn S, Gajewski J, Schulz J, Corcos J. A population-based study of urinary symptoms and incontinence: the Canadian Urinary Bladder Survey. BJU Int. 2008 Jan;101(1):52-8. doi: 10.1111/j.1464-410X.2007.07198.x. Epub 2007 Oct 1. PMID 17908260
- [Background] Almousa S, Bandin van Loon A. The prevalence of urinary incontinence in nulliparous adolescent and middle-aged women and the associated risk factors: A systematic review. Maturitas. 2018 Jan;107:78-83. doi: 10.1016/j.maturitas.2017.10.003. Epub 2017 Oct 7. PMID 29169586
- [Background] Windle G, Hughes D, Linck P, Russell I, Woods B. Is exercise effective in promoting mental well-being in older age? A systematic review. Aging Ment Health. 2010 Aug;14(6):652-69. doi: 10.1080/13607861003713232. PMID 20686977
- [Background] Sun F, Norman IJ, While AE. Physical activity in older people: a systematic review. BMC Public Health. 2013 May 6;13:449. doi: 10.1186/1471-2458-13-449. PMID 23648225
- [Background] Nygaard I, Girts T, Fultz NH, Kinchen K, Pohl G, Sternfeld B. Is urinary incontinence a barrier to exercise in women? Obstet Gynecol. 2005 Aug;106(2):307-14. doi: 10.1097/01.AOG.0000168455.39156.0f. PMID 16055580
- [Background] Smith AR, Hosker GL, Warrell DW. The role of pudendal nerve damage in the aetiology of genuine stress incontinence in women. Br J Obstet Gynaecol. 1989 Jan;96(1):29-32. doi: 10.1111/j.1471-0528.1989.tb01572.x. PMID 2923841
- [Background] Ree ML, Nygaard I, Bo K. Muscular fatigue in the pelvic floor muscles after strenuous physical activity. Acta Obstet Gynecol Scand. 2007;86(7):870-6. doi: 10.1080/00016340701417281. PMID 17611834
- [Background] Bo K. Urinary incontinence, pelvic floor dysfunction, exercise and sport. Sports Med. 2004;34(7):451-64. doi: 10.2165/00007256-200434070-00004. PMID 15233598
- [Background] Ashton-Miller JA, DeLancey JO. Functional anatomy of the female pelvic floor. Ann N Y Acad Sci. 2007 Apr;1101:266-96. doi: 10.1196/annals.1389.034. Epub 2007 Apr 7. PMID 17416924
- [Background] Dietz HP, Clarke B, Herbison P. Bladder neck mobility and urethral closure pressure as predictors of genuine stress incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2002;13(5):289-93. doi: 10.1007/s001920200063. PMID 12355287
- [Background] Rud T, Andersson KE, Asmussen M, Hunting A, Ulmsten U. Factors maintaining the intraurethral pressure in women. Invest Urol. 1980 Jan;17(4):343-7. PMID 7188694
- [Background] DeLancey JO. Structural support of the urethra as it relates to stress urinary incontinence: the hammock hypothesis. Am J Obstet Gynecol. 1994 Jun;170(6):1713-20; discussion 1720-3. doi: 10.1016/s0002-9378(94)70346-9. PMID 8203431
- [Background] DeLancey JO, Trowbridge ER, Miller JM, Morgan DM, Guire K, Fenner DE, Weadock WJ, Ashton-Miller JA. Stress urinary incontinence: relative importance of urethral support and urethral closure pressure. J Urol. 2008 Jun;179(6):2286-90; discussion 2290. doi: 10.1016/j.juro.2008.01.098. Epub 2008 Apr 18. PMID 18423707
- [Background] Pontbriand-Drolet S, Tang A, Madill SJ, Tannenbaum C, Lemieux MC, Corcos J, Dumoulin C. Differences in pelvic floor morphology between continent, stress urinary incontinent, and mixed urinary incontinent elderly women: An MRI study. Neurourol Urodyn. 2016 Apr;35(4):515-21. doi: 10.1002/nau.22743. Epub 2015 Mar 1. PMID 25727524
- [Background] Madill SJ, Harvey MA, McLean L. Women with SUI demonstrate motor control differences during voluntary pelvic floor muscle contractions. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Apr;20(4):447-59. doi: 10.1007/s00192-008-0800-y. Epub 2009 Jan 23. PMID 19165411
- [Background] Smith MD, Coppieters MW, Hodges PW. Postural activity of the pelvic floor muscles is delayed during rapid arm movements in women with stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Aug;18(8):901-11. doi: 10.1007/s00192-006-0259-7. Epub 2006 Dec 1. PMID 17139463
- [Background] Nygaard IE, Shaw JM. Physical activity and the pelvic floor. Am J Obstet Gynecol. 2016 Feb;214(2):164-171. doi: 10.1016/j.ajog.2015.08.067. Epub 2015 Sep 6. PMID 26348380
- [Background] Brandao S, Da Roza T, Mascarenhas T, Ramos I, Natal Jorge R. Do asymptomatic former high-impact sports practitioners maintain the ability to contract the pelvic floor muscles? J Sports Med Phys Fitness. 2015 Nov;55(11):1272-6. Epub 2014 Oct 30. PMID 25359130
- [Background] Varella LR, Torres VB, Angelo PH, Eugenia de Oliveira MC, Matias de Barros AC, Viana Ede S, Micussi MT. Influence of parity, type of delivery, and physical activity level on pelvic floor muscles in postmenopausal women. J Phys Ther Sci. 2016 Mar;28(3):824-30. doi: 10.1589/jpts.28.824. Epub 2016 Mar 31. PMID 27134366
- [Background] Bo K, Sherburn M. Evaluation of female pelvic-floor muscle function and strength. Phys Ther. 2005 Mar;85(3):269-82. PMID 15733051
- [Background] Middlekauff ML, Egger MJ, Nygaard IE, Shaw JM. The impact of acute and chronic strenuous exercise on pelvic floor muscle strength and support in nulliparous healthy women. Am J Obstet Gynecol. 2016 Sep;215(3):316.e1-7. doi: 10.1016/j.ajog.2016.02.031. Epub 2016 Feb 17. PMID 26899909
- [Background] Dumoulin C, Cacciari LP, Hay-Smith EJC. Pelvic floor muscle training versus no treatment, or inactive control treatments, for urinary incontinence in women. Cochrane Database Syst Rev. 2018 Oct 4;10(10):CD005654. doi: 10.1002/14651858.CD005654.pub4. PMID 30288727
- [Background] Ziv E, Stanton SL, Abarbanel J. Efficacy and safety of a novel disposable intravaginal device for treating stress urinary incontinence. Am J Obstet Gynecol. 2008 May;198(5):594.e1-7. doi: 10.1016/j.ajog.2008.01.061. Epub 2008 Apr 2. PMID 18377862
- [Background] Ziv E, Stanton SL, Abarbanel J. Significant improvement in the quality of life in women treated with a novel disposable intravaginal device for stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Jun;20(6):651-8. doi: 10.1007/s00192-009-0824-y. Epub 2009 Mar 11. PMID 19434384
- [Background] Milne JL, Robert M, Tang S, Drummond N, Ross S. Goal achievement as a patient-generated outcome measure for stress urinary incontinence. Health Expect. 2009 Sep;12(3):288-300. doi: 10.1111/j.1369-7625.2009.00536.x. PMID 19754692
- [Background] Melin A, Tornberg AB, Skouby S, Faber J, Ritz C, Sjodin A, Sundgot-Borgen J. The LEAF questionnaire: a screening tool for the identification of female athletes at risk for the female athlete triad. Br J Sports Med. 2014 Apr;48(7):540-5. doi: 10.1136/bjsports-2013-093240. Epub 2014 Feb 21. PMID 24563388
- [Background] Hagstromer M, Oja P, Sjostrom M. The International Physical Activity Questionnaire (IPAQ): a study of concurrent and construct validity. Public Health Nutr. 2006 Sep;9(6):755-62. doi: 10.1079/phn2005898. PMID 16925881
- [Background] Bo K. Reproducibility of instruments designed to measure subjective evaluation of female stress urinary incontinence. Scand J Urol Nephrol. 1994 Mar;28(1):97-100. doi: 10.3109/00365599409180479. PMID 8009197
- [Background] Berube ME, Czyrnyj CS, McLean L. An automated intravaginal dynamometer: Reliability metrics and the impact of testing protocol on active and passive forces measured from the pelvic floor muscles. Neurourol Urodyn. 2018 Aug;37(6):1875-1888. doi: 10.1002/nau.23575. Epub 2018 Apr 10. PMID 29635776
- [Background] Thibault-Gagnon S, Gentilcore-Saulnier E, Auchincloss C, McLean L. Pelvic floor ultrasound imaging: are physiotherapists interchangeable in the assessment of levator hiatal biometry? Physiother Can. 2014 Fall;66(4):340-7. doi: 10.3138/ptc.2013-50. PMID 25922555
- [Background] Braekken IH, Majida M, Ellstrom-Engh M, Dietz HP, Umek W, Bo K. Test-retest and intra-observer repeatability of two-, three- and four-dimensional perineal ultrasound of pelvic floor muscle anatomy and function. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Feb;19(2):227-35. doi: 10.1007/s00192-007-0408-7. Epub 2007 Jun 29. PMID 17599234
- [Background] Braekken IH, Majida M, Engh ME, Bo K. Test-retest reliability of pelvic floor muscle contraction measured by 4D ultrasound. Neurourol Urodyn. 2009;28(1):68-73. doi: 10.1002/nau.20618. PMID 18932174
- [Background] Burgio KL, Goode PS, Richter HE, Locher JL, Roth DL. Global ratings of patient satisfaction and perceptions of improvement with treatment for urinary incontinence: validation of three global patient ratings. Neurourol Urodyn. 2006;25(5):411-7. doi: 10.1002/nau.20243. PMID 16652380
- [Derived] Vesting S, Petter Rodrigues M, Collins G, McLean L. Intravaginal devices for running-induced urinary incontinence symptoms in females: a study protocol. BJU Int. 2025 Jun;135(6):931-939. doi: 10.1111/bju.16708. Epub 2025 Mar 12. PMID 40071535